CLINICAL TRIAL: NCT03691610
Title: Immunogenicity and Safety Study of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers
Brief Title: Immunogenicity and Safety Study of a Quadrivalent Meningococcal Conjugate Vaccine Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET61; U1111-1205-2836 (Registry Identifier: ICTRP); MET61 (Other: Sanofi Identifier); 2019-004460-22 (EudraCT Number)
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers (Meningococcal Infection)
MeSH Terms: conditions — Meningococcal Infections | interventions — Tetanus Toxoid; HibTITER protein, Haemophilus influenzae; Hepatitis B Vaccines; Poliovirus Vaccine, Inactivated; 13-valent pneumococcal vaccine; Rotavirus Vaccines; Measles-Mumps-Rubella Vaccine; Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study has a modified double blind design for each group at enrollment, and thus, with the exception of the personnel administering the vaccine, everyone involved in study is blinded to avoid any bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): MenACYW conjugate vaccine + routine pediatric vaccines at 6 to 7 months of age and 12 to 13 months of age
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A,C,Y and W) Tetanus Toxoid Conjugate vaccine MenACYW conjugate vaccine; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis, inactivated Poliovirus and Haemophilus b Conjugate Vaccine; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis, Hepatitis B and Inactivated Poliovirus Vaccine; Biological: Haemophilus b Conjugate Vaccine; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Hepatitis B Vaccine; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live
- Group 2 (Active Comparator): MENVEO® + routine pediatric vaccines at 6 to 7 months of age and 12 to 13 months of age
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis, inactivated Poliovirus and Haemophilus b Conjugate Vaccine; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis, Hepatitis B and Inactivated Poliovirus Vaccine; Biological: Haemophilus b Conjugate Vaccine; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Hepatitis B Vaccine; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Varicella Virus Vaccine Live
- Group 3 (Experimental): MenACYW conjugate vaccine at 17 to 19 months of age and 20 to 23 months of age
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A,C,Y and W) Tetanus Toxoid Conjugate vaccine MenACYW conjugate vaccine
- Group 4 (Active Comparator): Menactra® at 17 to 19 months of age and 20 to 23 months of age
  Interventions: Biological: Meningococcal Polysaccharide (serogroups A,C,Y and W-135) Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A,C,Y and W) Tetanus Toxoid Conjugate vaccine MenACYW conjugate vaccine — Pharmaceutical form:Solution for injection Route of administration: Intramuscular, 0.5 mL
  Arms: Group 1; Group 3
Biological: Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine — Pharmaceutical form: Solution for injection Route of administration: Intramuscular, 0.5 mL
  Arms: Group 2
Biological: Meningococcal Polysaccharide (serogroups A,C,Y and W-135) Diphtheria Toxoid Conjugate Vaccine — Pharmaceutical form: Solution for injection Route of administration: Intramuscular, 0.5 mL
  Arms: Group 4
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis, inactivated Poliovirus and Haemophilus b Conjugate Vaccine — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular, 0.5 mL
  Arms: Group 1; Group 2
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis, Hepatitis B and Inactivated Poliovirus Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular, 0.5 mL
  Arms: Group 1; Group 2
Biological: Haemophilus b Conjugate Vaccine — Pharmaceutical form:Solution for injection Route of administration: Intramuscular, 0.5 mL
  Arms: Group 1; Group 2
Biological: Pneumococcal 13-valent Conjugate Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular, 0.5 mL
  Arms: Group 1; Group 2
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — Pharmaceutical form:Oral solution Route of administration: Oral, 2 mL
  Arms: Group 1; Group 2
Biological: Hepatitis B Vaccine — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular, 0.5 mL
  Arms: Group 1; Group 2
Biological: Measles, Mumps, and Rubella Virus Vaccine Live — Pharmaceutical form: Lyophilized live virus vaccine Route of administration: Subcutaneous, 0.5 mL
  Arms: Group 1; Group 2
Biological: Varicella Virus Vaccine Live — Pharmaceutical form:Suspension for injection Route of administration: Subcutaneous, 0.5 mL
  Arms: Group 1; Group 2

SUMMARY:
The primary objective of this study is to demonstrate the non-inferiority of the vaccine seroresponse to meningococcal serogroups A, C, Y, and W following administration of 2 doses of MenACYW conjugate vaccine compared to 2 doses of MENVEO® when given concomitantly with routine pediatric vaccines to infants and toddlers 6 to 7 months of age and 12 to 13 months of age.

The secondary objectives of the study are:

* To demonstrate the non-inferiority of the percentage of participants with antibody titers to meningococcal serogroups A, C, Y, and W ≥ 1:8 following administration of 2 doses of MenACYW conjugate vaccine compared to 2 doses of MENVEO® when given concomitantly with pediatric routine vaccines to infants and toddlers at 6 to 7 months of age and 12 to 13 months of age.
* To describe the antibody response against meningococcal serogroups A, C, Y, and W 30 days after the second vaccination at 12 to 13 months of age with MenACYW conjugate vaccine or MENVEO®.
* To describe the antibody response against meningococcal serogroups A, C, Y, and W 30 days and 6 months after the first vaccination at 6 to 7 months of age with MenACYW conjugate vaccine or MENVEO®.
* To describe the antibody response against meningococcal serogroups A, C, Y, and W 30 days after the second vaccination at 20 to 23 months of age with MenACYW conjugate vaccine or Menactra®.

DETAILED DESCRIPTION:
Study duration per participant is approximately 1 year in Group 1 and Group 2, and 10 months in Group 3 and Group 4. This duration includes a safety follow-up contact at 6 months after the last vaccination.

ELIGIBILITY:
Inclusion criteria :

* Aged 6 to 7 months (168 to 224 days) or 17 to 19 months on the day of the first visit
* Informed consent form has been signed and dated by the parent(s) or other guardian and by an independent witness if required by local regulations
* Subject and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures
* For subjects 6 to 7 months of age at enrollment (Group 1 and Group 2), documented history of having received 2 doses of diphtheria, tetanus and acellular pertussis (DTaP), Haemophilus influenza type B (Hib), inactivated poliovirus (IPV), pneumococcal, hepatitis B (for children who received hepatitis B at 2 and 4 months of age, prior receipt of 3 doses of hepatitis B), and rotavirus vaccines
* For subjects to be enrolled at 17 to 19 months of age (Group 3 and Group 4), documented history of having received all routine pediatric vaccines recommended by the Advisory Committee on Immunization Practices (ACIP) up to the age of enrollment

Exclusion criteria:

* Participation at the time of study enrollment or in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks before and / or following any trial vaccination except for influenza vaccination, which may be received at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B serogroup-containing vaccine)
* For subjects to be enrolled at 6 to 7 months of age (Group 1 and Group 2), prior receipt of more than 2 doses of rotavirus vaccine (Rotateq), DTaP, Hib, IPV, pneumococcal, hepatitis B (for children who received hepatitis B at 2 and 4 months of age, prior receipt of more than 3 doses of hepatitis B vaccine)
* For subjects to be enrolled at 6 to 7 months of age (Group 1 and Group 2), receipt of the 2 doses of rotavirus vaccine at 2 and 4 months of age
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) within the past 3 months
* Family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated
* Individuals with blood dyscrasias, leukemia, lymphoma of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems
* Individuals with active tuberculosis
* History of any Neisseria meningitidis infection, confirmed either clinically, serologically, or microbiologically
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, hepatitis A, measles, mumps, rubella, varicella; and of Haemophilus influenzae type b, Streptococcus pneumoniae, and /or rotavirus infection or disease
* At high risk for meningococcal infection during the trial (specifically, but not limited to, subjects with persistent complement deficiency, with anatomic or functional asplenia, or subjects travelling to countries with high endemic or epidemic disease)
* History of intussusception
* History of any neurologic disorders, including any seizures and progressive neurologic disorders
* History of Arthus-type hypersensitivity reaction after a previous dose of tetanus toxoid-containing vaccine
* History of Guillain-Barré syndrome
* Known systemic hypersensitivity to any of the vaccine components or to latex, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances, including neomycin, gelatin, and yeast
* Verbal report of thrombocytopenia contraindicating intramuscular vaccination in the investigator's opinion
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the investigator's opinion
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0 C [≥ 100.4 F]). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as a natural or adopted child of the investigator or employee with direct involvement in the proposed study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 950 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (47):
- United States (45):
  - Alabama Clinical Therapeutics Site Number : 8400036, Birmingham, Alabama
  - Southeastern Pediatric Associates Site Number : 8400009, Dothan, Alabama
  - MedPharmics, LLC - Phoenix Site Number : 8400013, Phoenix, Arizona
  - Emmaus Research Center, Inc Site Number : 8400019, Anaheim, California
  - Coast Clinical Trials, LLC Site Number : 8400073, Bellflower, California
  - Matrix Clinical Research Site Number : 8400082, Gardena, California
  - Madera Family Med Group Site Number : 8400065, Madera, California
  - Next Phase Research Alliance Site Number : 8400044, Homestead, Florida
  - PAS Research Site Number : 8400101, Land O' Lakes, Florida
  - Axcess Medical Research Site Number : 8400021, Loxahatchee Groves, Florida
  - Y and L Advance Health Care, Inc D/B/A Elite Clinical Res Site Number : 8400046, Miami, Florida
  - Biomedical Research LLC Site Number : 8400041, Miami, Florida
  - Crystal Biomedical Research Site Number : 8400034, Miami Lakes, Florida
  - PAS Research Site Number : 8400059, Tampa, Florida
  - Omega Pediatrics Site Number : 8400093, Roswell, Georgia
  - Snake River Research, PLLC Site Number : 8400058, Idaho Falls, Idaho
  - Eagle Clinical Research Site Number : 8400094, Chicago, Illinois
  - Brownsboro Park Pediatrics Site Number : 8400039, Louisville, Kentucky
  - All Children Pediatrics Site Number : 8400024, Louisville, Kentucky
  - Meridian Clinical Research, LLC Site Number : 8400035, Baton Rouge, Louisiana
  - Velocity Clinical Research Site Number : 8400016, Metairie, Louisiana
  - Willis-Knighton Physician Network Site Number : 8400075, Shreveport, Louisiana
  - Victory Clinical Research Site Number : 8400026, Baltimore, Maryland
  - Pediatric Associates of Fall River Site Number : 8400112, Fall River, Massachusetts
  - Craig Spiegel, MD Site Number : 8400023, Bridgeton, Missouri
  - Meridian Clinical Research Site Number : 8400097, Hastings, Nebraska
  - Midwest Childrens Health Research Institute Site Number : 8400111, Lincoln, Nebraska
  - Midwest Childrens Health Research Institute Site Number : 8400117, Lincoln, Nebraska
  - MedPharmics Inc Site Number : 8400006, Albuquerque, New Mexico
  - Advantage Clinical Trials Site Number : 8400069, New York, New York
  - Wilmington Health Site Number : 8400054, Wilmington, North Carolina
  - Ohio Pediatric Research Site Number : 8400022, Dayton, Ohio
  - PriMed Clinical Research Site Number : 8400008, Dayton, Ohio
  - Oklahoma State University - Center for Health Sciences Site Number : 8400110, Tulsa, Oklahoma
  - Cyn3rgy Research Site Number : 8400010, Gresham, Oregon
  - Allegheny Health and Wellness Pavilion Site Number : 8400025, Erie, Pennsylvania
  - Kid's Way Pediatrics Site Number : 8400015, Hermitage, Pennsylvania
  - Coastal Pediatric Research Charleston Site Number : 8400002, Charleston, South Carolina
  - Coastal Pediatric Research Charleston Site Number : 8400011, Charleston, South Carolina
  - Tribe Clinical Research Site Number : 8400118, Greenville, South Carolina
  - Pediatric Clinical Trials Tullahoma Site Number : 8400106, Tullahoma, Tennessee
  - Tekton Research Site Number : 8400047, Beaumont, Texas
  - Mercury Clinical Research, Inc. Site Number : 8400088, Dickinson, Texas
  - Clinical Trial Network - 7080 Southwest Fwy Site Number : 8400037, Houston, Texas
  - Tekton Research, Inc. Site Number : 8400040, San Antonio, Texas
- Puerto Rico (2):
  - Investigational Site Number : 6300102, Guayama
  - Investigational Site Number : 6300014, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 47 centers in the United States and Puerto Rico between 04 October 2018 and 23 October 2023.
Pre-assignment Details: A total of 950 participants were enrolled and randomized in the study.
Groups:
- Infants: Group 1: Participants received 2 doses of meningococcal polysaccharide (serogroups A, C, Y and W [MenACYW conjugate vaccine]) 0.5 milliliter (mL) intramuscular (IM) injection at 6 to 7 month of age (MoA) and 12 to 13 MoA, co-administered with pediatric vaccines recommended at this age.
- Infants: Group 2: Participants received 2 doses of MENVEO® 0.5 mL IM injection at 6 to 7 MoA and 12 to 13 MoA, co-administered with pediatric vaccines recommended at this age.
- Toddlers: Group 3: Participants received 2 doses of meningococcal polysaccharide (serogroups A, C, Y and W [MenACYW conjugate vaccine]) 0.5 mL IM injection at 17 to 19 MoA and 20 to 23 MoA.
- Toddlers: Group 4: Participants received 2 doses of Menactra® 0.5 mL IM injection at 17 to 19 MoA and 20 to 23 MoA.
Period: Overall Study
Arm/Group | Infants: Group 1 | Infants: Group 2 | Toddlers: Group 3 | Toddlers: Group 4
Started | 380 | 370 | 96 | 104
Completed | 298 | 290 | 83 | 94
Not Completed | 82 | 80 | 13 | 10
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 15 | 8 | 1 | 2
Not completed — Withdrawal by Parent/Guardian | 47 | 60 | 7 | 6
Not completed — Lost to Follow-up | 20 | 11 | 5 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of the study vaccine.
Groups:
- Infants: Group 1: Participants received 2 doses of meningococcal polysaccharide (serogroups A, C, Y and W [MenACYW conjugate vaccine]) 0.5 mL IM injection at 6 to 7 MoA and 12 to 13 MoA, co-administered with pediatric vaccines recommended at this age.
- Total: Total of all reporting groups
Arm/Group | Infants: Group 1 | Infants: Group 2 | Toddlers: Group 3 | Toddlers: Group 4 | Total
Number analyzed (Participants) | 380 | 370 | 96 | 104 | 950
Age, Continuous [Mean (Standard Deviation); unit: Units: months] — Population: One participant in 'Infants: Group 1' reporting group had missing value of age.
  Units: months
    number analyzed (Participants) | 379 | 370 | 96 | 104 | 949
    (all) | 6.01 (0.700) | 6.02 (0.396) | 17.9 (0.632) | 17.9 (0.673) | 8.51 (4.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 172 | 48 | 52 | 452
  Male | 200 | 198 | 48 | 52 | 498
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 6 | 6 | 2 | 1 | 15
  Black or African American | 70 | 68 | 11 | 11 | 160
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 277 | 264 | 79 | 87 | 707
  Mixed origin | 14 | 20 | 4 | 5 | 43
  Not Reported | 10 | 4 | 0 | 0 | 14
  Unknown | 3 | 7 | 0 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Infants Groups 1 and 2: Percentage of Participants With Vaccine Seroresponse Measured by Serum Bactericidal Assay Using Human Complement (hSBA) at 30 Days Post Second Dose of MenACYW Conjugate Vaccine or MENVEO
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. The hSBA vaccine seroresponse was defined as a post-vaccination titer >= 1:16 for participants with pre-vaccination hSBA titer < 1:8, or a post-vaccination titer >= 4-fold increase from baseline for participant with pre-vaccination hSBA titer >= 1:8.
Time Frame: Baseline (Day 0) and 30 days post second dose (12 to 13 MoA) of MenACYW conjugate vaccine or MENVEO, maximum of 14 months
Population: Per-protocol analysis set 2 (PPAS2) was a subset of the full analysis set 2 (FAS2). The FAS2 included all randomized participants who received at least 1 dose of the study vaccine in the second year of life (>= 12 MOA) and had a valid post vaccination serology result in the second year of life. Only participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infants: Group 1 | Infants: Group 2
Number analyzed (Participants) | 143 | 128
percentage of participants
  Serogroup A: number analyzed (Participants) | 141 | 123
  Serogroup A | 89.4 [83.1 to 93.9] | 82.9 [75.1 to 89.1]
  Serogroup C: number analyzed (Participants) | 134 | 126
  Serogroup C | 99.3 [95.9 to 100] | 97.6 [93.2 to 99.5]
  Serogroup Y: number analyzed (Participants) | 140 | 128
  Serogroup Y | 98.6 [94.9 to 99.8] | 97.7 [93.3 to 99.5]
  Serogroup W: number analyzed (Participants) | 143 | 127
  Serogroup W | 99.3 [96.2 to 100] | 92.9 [87.0 to 96.7]

2. Secondary Outcome: Infants Groups 1 and 2: Percentage of Participants Who Achieved Antibody Titer (Seroprotection) >=1:8 by hSBA at 30 Days Post Second Dose of MenACYW Conjugate Vaccine or MENVEO
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. Seroprotection rate was defined as percentage of participants with hSBA titers >= 1:8.
Time Frame: At 30 days post second dose (12 to 13 MoA) of MenACYW conjugate vaccine or MENVEO
Population: The PPAS2 was a subset of the FAS2. The FAS2 included all randomized participants who received at least 1 dose of the study vaccine in the second year of life (>= 12 MOA) and had a valid post vaccination serology result in the second year of life. Only participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infants: Group 1 | Infants: Group 2
Number analyzed (Participants) | 171 | 160
percentage of participants
  Serogroup A: number analyzed (Participants) | 170 | 158
  Serogroup A | 95.3 [90.9 to 97.9] | 93.0 [87.9 to 96.5]
  Serogroup C: number analyzed (Participants) | 162 | 160
  Serogroup C | 100 [97.7 to 100] | 98.1 [94.6 to 99.6]
  Serogroup Y: number analyzed (Participants) | 170 | 160
  Serogroup Y | 100 [97.9 to 100] | 97.5 [93.7 to 99.3]
  Serogroup W: number analyzed (Participants) | 171 | 159
  Serogroup W | 100 [97.9 to 100] | 95.6 [91.1 to 98.2]

3. Secondary Outcome: Infants Groups 1 and 2: Percentage of Participants With hSBA Antibody Titer >= 1:4 and >= 1:8
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. Participants with hSBA titers >= 1:4 and >= 1:8 were analyzed. PPAS1= Per-Protocol Analysis Set 1; FAS1= Full analysis set 1; PPAS3= Per-Protocol Analysis Set 3; and FAS3= Full analysis set 3.
Time Frame: PPAS1: At 30 days post first dose (6 to 7 MoA); PPAS2: At Baseline (pre-dose on Day 0) and 30 days post second dose (12 to 13 MoA); and PPAS3: At 6 months post first dose (6 to 7 MoA) of MenACYW conjugate vaccine or MENVEO
Population: PPAS1 was a subset of FAS1. FAS1 included all randomized participants who received at least 1 dose of study vaccine in infancy (< 12 MOA) and had a valid post vaccination serology result in infancy. PPAS2 analysis set. PPAS3 was a subset of FAS3. FAS3 included all randomized participants who received at least 1 dose of study vaccine in infancy and had a valid pre-vaccination serology result at visit 3. Only participants with data collected for each serogroup at specific timepoint are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infants: Group 1 | Infants: Group 2
Number analyzed (Participants) | 171 | 160
percentage of participants
  PPAS1, Serogroup A: >=1:4: number analyzed (Participants) | 130 | 132
  PPAS1, Serogroup A: >=1:4 | 64.6 [55.8 to 72.8] | 55.3 [46.4 to 64.0]
  PPAS1, Serogroup A: >=1:8: number analyzed (Participants) | 130 | 132
  PPAS1, Serogroup A: >=1:8 | 54.6 [45.7 to 63.4] | 37.9 [29.6 to 46.7]
  PPAS1, Serogroup C: >=1:4: number analyzed (Participants) | 127 | 133
  PPAS1, Serogroup C: >=1:4 | 96.9 [92.1 to 99.1] | 93.2 [87.5 to 96.9]
  PPAS1, Serogroup C: >=1:8: number analyzed (Participants) | 127 | 133
  PPAS1, Serogroup C: >=1:8 | 96.9 [92.1 to 99.1] | 90.2 [83.9 to 94.7]
  PPAS1, Serogroup Y: >=1:4: number analyzed (Participants) | 125 | 128
  PPAS1, Serogroup Y: >=1:4 | 70.4 [61.6 to 78.2] | 43.0 [34.3 to 52.0]
  PPAS1, Serogroup Y: >=1:8: number analyzed (Participants) | 125 | 128
  PPAS1, Serogroup Y: >=1:8 | 60.8 [51.7 to 69.4] | 26.6 [19.1 to 35.1]
  PPAS1, Serogroup W: >=1:4: number analyzed (Participants) | 134 | 134
  PPAS1, Serogroup W: >=1:4 | 49.3 [40.5 to 58.0] | 37.3 [29.1 to 46.1]
  PPAS1, Serogroup W: >=1:8: number analyzed (Participants) | 134 | 134
  PPAS1, Serogroup W: >=1:8 | 38.1 [29.8 to 46.8] | 28.4 [20.9 to 36.8]
  PPAS2, Serogroup A, Day 0: >=1:4: number analyzed (Participants) | 144 | 127
  PPAS2, Serogroup A, Day 0: >=1:4 | 56.3 [47.7 to 64.5] | 51.2 [42.2 to 60.1]
  PPAS2, Serogroup A, Day 0: >=1:8: number analyzed (Participants) | 144 | 127
  PPAS2, Serogroup A, Day 0: >=1:8 | 29.2 [21.9 to 37.3] | 24.4 [17.2 to 32.8]
  PPAS2, Serogroup A, Day 30: >=1:4: number analyzed (Participants) | 170 | 158
  PPAS2, Serogroup A, Day 30: >=1:4 | 97.1 [93.3 to 99.0] | 94.9 [90.3 to 97.8]
  PPAS2, Serogroup A, Day 30: >=1:8: number analyzed (Participants) | 170 | 158
  PPAS2, Serogroup A, Day 30: >=1:8 | 95.3 [90.9 to 97.9] | 93.0 [87.9 to 96.5]
  PPAS2, Serogroup C, Day 0: >=1:4: number analyzed (Participants) | 147 | 129
  PPAS2, Serogroup C, Day 0: >=1:4 | 10.2 [5.8 to 16.3] | 12.4 [7.3 to 19.4]
  PPAS2, Serogroup C, Day 0: >=1:8: number analyzed (Participants) | 147 | 129
  PPAS2, Serogroup C, Day 0: >=1:8 | 6.1 [2.8 to 11.3] | 7.0 [3.2 to 12.8]
  PPAS2, Serogroup C, Day 30: >=1:4: number analyzed (Participants) | 162 | 160
  PPAS2, Serogroup C, Day 30: >=1:4 | 100 [97.7 to 100] | 99.4 [96.6 to 100]
  PPAS2, Serogroup C, Day 30: >=1:8: number analyzed (Participants) | 162 | 160
  PPAS2, Serogroup C, Day 30: >=1:8 | 100 [97.7 to 100] | 98.1 [94.6 to 99.6]
  PPAS2, Serogroup Y, Day 0: >=1:4: number analyzed (Participants) | 149 | 130
  PPAS2, Serogroup Y, Day 0: >=1:4 | 15.4 [10.0 to 22.3] | 12.3 [7.2 to 19.2]
  PPAS2, Serogroup Y, Day 0: >=1:8: number analyzed (Participants) | 149 | 130
  PPAS2, Serogroup Y, Day 0: >=1:8 | 8.7 [4.7 to 14.5] | 6.2 [2.7 to 11.8]
  PPAS2, Serogroup Y, Day 30: >=1:4: number analyzed (Participants) | 170 | 160
  PPAS2, Serogroup Y, Day 30: >=1:4 | 100 [97.9 to 100] | 98.1 [94.6 to 99.6]
  PPAS2, Serogroup Y, Day 30: >=1:8: number analyzed (Participants) | 170 | 160
  PPAS2, Serogroup Y, Day 30: >=1:8 | 100 [97.9 to 100] | 97.5 [93.7 to 99.3]
  PPAS2, Serogroup W, Day 0: >=1:4: number analyzed (Participants) | 148 | 130
  PPAS2, Serogroup W, Day 0: >=1:4 | 6.8 [3.3 to 12.1] | 10.8 [6.0 to 17.4]
  PPAS2, Serogroup W, Day 0: >=1:8: number analyzed (Participants) | 148 | 130
  PPAS2, Serogroup W, Day 0: >=1:8 | 4.7 [1.9 to 9.5] | 6.2 [2.7 to 11.8]
  PPAS2, Serogroup W, Day 30: >=1:4: number analyzed (Participants) | 171 | 159
  PPAS2, Serogroup W, Day 30: >=1:4 | 100 [97.9 to 100] | 96.9 [92.8 to 99.0]
  PPAS2, Serogroup W, Day 30: >=1:8: number analyzed (Participants) | 171 | 159
  PPAS2, Serogroup W, Day 30: >=1:8 | 100 [97.9 to 100] | 95.6 [91.1 to 98.2]
  PPAS3, Serogroup A: >=1:4: number analyzed (Participants) | 103 | 91
  PPAS3, Serogroup A: >=1:4 | 87.4 [79.4 to 93.1] | 85.7 [76.8 to 92.2]
  PPAS3, Serogroup A: >=1:8: number analyzed (Participants) | 103 | 91
  PPAS3, Serogroup A: >=1:8 | 77.7 [68.4 to 85.3] | 73.6 [63.3 to 82.3]
  PPAS3, Serogroup C: >=1:4: number analyzed (Participants) | 104 | 94
  PPAS3, Serogroup C: >=1:4 | 99.0 [94.8 to 100] | 77.7 [67.9 to 85.6]
  PPAS3, Serogroup C: >=1:8: number analyzed (Participants) | 104 | 94
  PPAS3, Serogroup C: >=1:8 | 98.1 [93.2 to 99.8] | 69.1 [58.8 to 78.3]
  PPAS3, Serogroup Y: >=1:4: number analyzed (Participants) | 106 | 93
  PPAS3, Serogroup Y: >=1:4 | 98.1 [93.4 to 99.8] | 69.9 [59.5 to 79.0]
  PPAS3, Serogroup Y: >=1:8: number analyzed (Participants) | 106 | 93
  PPAS3, Serogroup Y: >=1:8 | 96.2 [90.6 to 99.0] | 54.8 [44.2 to 65.2]
  PPAS3, Serogroup W: >=1:4: number analyzed (Participants) | 106 | 93
  PPAS3, Serogroup W: >=1:4 | 98.1 [93.4 to 99.8] | 61.3 [50.6 to 71.2]
  PPAS3, Serogroup W: >=1:8: number analyzed (Participants) | 106 | 93
  PPAS3, Serogroup W: >=1:8 | 96.2 [90.6 to 99.0] | 50.5 [40.0 to 61.1]

4. Secondary Outcome: Infants Groups 1 and 2: Geometric Mean Titers Against Meningococcal Serogroups A, C, W, and Y
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA and the results were expressed as geometric mean titers.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Infants: Group 1 | Infants: Group 2
Number analyzed (Participants) | 171 | 160
titer
  PPAS1: Serogroup A: number analyzed (Participants) | 130 | 132
  PPAS1: Serogroup A | 8.26 [6.55 to 10.4] | 5.45 [4.42 to 6.72]
  PPAS1: Serogroup C: number analyzed (Participants) | 127 | 133
  PPAS1: Serogroup C | 167 [129 to 217] | 41.3 [32.8 to 52.1]
  PPAS1: Serogroup Y: number analyzed (Participants) | 125 | 128
  PPAS1: Serogroup Y | 8.36 [6.61 to 10.6] | 3.79 [3.20 to 4.49]
  PPAS1: Serogroup W: number analyzed (Participants) | 134 | 134
  PPAS1: Serogroup W | 5.51 [4.39 to 6.92] | 3.82 [3.22 to 4.52]
  PPAS2, Serogroup A: Day 0: number analyzed (Participants) | 144 | 127
  PPAS2, Serogroup A: Day 0 | 4.73 [3.92 to 5.72] | 4.64 [3.74 to 5.74]
  PPAS2, Serogroup A: Day 30: number analyzed (Participants) | 170 | 158
  PPAS2, Serogroup A: Day 30 | 184 [143 to 237] | 119 [90.6 to 157]
  PPAS2, Serogroup C: Day 0: number analyzed (Participants) | 147 | 129
  PPAS2, Serogroup C: Day 0 | 2.57 [2.21 to 2.99] | 2.48 [2.20 to 2.79]
  PPAS2, Serogroup C: Day 30: number analyzed (Participants) | 162 | 160
  PPAS2, Serogroup C: Day 30 | 1473 [1236 to 1756] | 319 [263 to 388]
  PPAS2, Serogroup Y: Day 0: number analyzed (Participants) | 149 | 130
  PPAS2, Serogroup Y: Day 0 | 2.54 [2.27 to 2.83] | 2.37 [2.16 to 2.60]
  PPAS2, Serogroup Y: Day 30: number analyzed (Participants) | 170 | 160
  PPAS2, Serogroup Y: Day 30 | 423 [358 to 499] | 133 [107 to 166]
  PPAS2, Serogroup W: Day 0: number analyzed (Participants) | 148 | 130
  PPAS2, Serogroup W: Day 0 | 2.23 [2.05 to 2.42] | 2.31 [2.13 to 2.51]
  PPAS2, Serogroup W: Day 30: number analyzed (Participants) | 171 | 159
  PPAS2, Serogroup W: Day 30 | 442 [367 to 533] | 106 [83.4 to 135]
  PPAS3: Serogroup A: number analyzed (Participants) | 103 | 91
  PPAS3: Serogroup A | 20.1 [14.7 to 27.4] | 14.9 [11.0 to 20.3]
  PPAS3: Serogroup C: number analyzed (Participants) | 104 | 94
  PPAS3: Serogroup C | 150 [117 to 193] | 12.7 [9.63 to 16.8]
  PPAS3: Serogroup Y: number analyzed (Participants) | 106 | 93
  PPAS3: Serogroup Y | 46.2 [36.3 to 58.6] | 6.74 [5.43 to 8.36]
  PPAS3: Serogroup W: number analyzed (Participants) | 106 | 93
  PPAS3: Serogroup W | 46.8 [36.1 to 60.5] | 6.16 [4.87 to 7.80]

5. Secondary Outcome: Infants Groups 1 and 2: Percentage of Participants With hSBA Antibody Titer >=1:4 to >= 1:128
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. Participants with hSBA titers >= 1:4 to >= 1:128 were analyzed.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Infants: Group 1 | Infants: Group 2
Number analyzed (Participants) | 171 | 160
percentage of participants
  PPAS1, Serogroup A: >=1:4: number analyzed (Participants) | 130 | 132
  PPAS1, Serogroup A: >=1:4 | 64.6 | 55.3
  PPAS1, Serogroup A: >=1:128: number analyzed (Participants) | 130 | 132
  PPAS1, Serogroup A: >=1:128 | 3.1 | 3.0
  PPAS1, Serogroup C: >=1:4: number analyzed (Participants) | 127 | 133
  PPAS1, Serogroup C: >=1:4 | 96.9 | 93.2
  PPAS1, Serogroup C: >=1:128: number analyzed (Participants) | 127 | 133
  PPAS1, Serogroup C: >=1:128 | 67.7 | 32.3
  PPAS1, Serogroup Y: >=1:4: number analyzed (Participants) | 125 | 128
  PPAS1, Serogroup Y: >=1:4 | 70.4 | 43.0
  PPAS1, Serogroup Y: >=1:128: number analyzed (Participants) | 125 | 128
  PPAS1, Serogroup Y: >=1:128 | 5.6 | 0.8
  PPAS1, Serogroup W: >=1:4: number analyzed (Participants) | 134 | 134
  PPAS1, Serogroup W: >=1:4 | 49.3 | 37.3
  PPAS1, Serogroup W: >=1:128: number analyzed (Participants) | 134 | 134
  PPAS1, Serogroup W: >=1:128 | 4.5 | 0
  PPAS2, Serogroup A, Day 0: >=1:4: number analyzed (Participants) | 144 | 127
  PPAS2, Serogroup A, Day 0: >=1:4 | 56.3 | 51.2
  PPAS2, Serogroup A, Day 0: >=1:128: number analyzed (Participants) | 144 | 127
  PPAS2, Serogroup A, Day 0: >=1:128 | 4.9 | 3.1
  PPAS2, Serogroup A, Day 30: >=1:4: number analyzed (Participants) | 170 | 158
  PPAS2, Serogroup A, Day 30: >=1:4 | 97.1 | 94.9
  PPAS2, Serogroup A, Day 30: >=1:128: number analyzed (Participants) | 170 | 158
  PPAS2, Serogroup A, Day 30: >=1:128 | 68.8 | 62.7
  PPAS2, Serogroup C, Day 0: >=1:4: number analyzed (Participants) | 147 | 129
  PPAS2, Serogroup C, Day 0: >=1:4 | 10.2 | 12.4
  PPAS2, Serogroup C, Day 0: >=1:128: number analyzed (Participants) | 147 | 129
  PPAS2, Serogroup C, Day 0: >=1:128 | 2.0 | 0
  PPAS2, Serogroup C, Day 30: >=1:4: number analyzed (Participants) | 162 | 160
  PPAS2, Serogroup C, Day 30: >=1:4 | 100 | 99.4
  PPAS2, Serogroup C, Day 30: >=1:128: number analyzed (Participants) | 162 | 160
  PPAS2, Serogroup C, Day 30: >=1:128 | 98.1 | 88.1
  PPAS2, Serogroup Y, Day 0: >=1:4: number analyzed (Participants) | 149 | 130
  PPAS2, Serogroup Y, Day 0: >=1:4 | 15.4 | 12.3
  PPAS2, Serogroup Y, Day 0: >=1:128: number analyzed (Participants) | 149 | 130
  PPAS2, Serogroup Y, Day 0: >=1:128 | 0.7 | 0
  PPAS2, Serogroup Y, Day 30: >=1:4: number analyzed (Participants) | 170 | 160
  PPAS2, Serogroup Y, Day 30: >=1:4 | 100 | 98.1
  PPAS2, Serogroup Y, Day 30: >=1:128: number analyzed (Participants) | 170 | 160
  PPAS2, Serogroup Y, Day 30: >=1:128 | 90.0 | 58.8
  PPAS2, Serogroup W, Day 0: >=1:4: number analyzed (Participants) | 148 | 130
  PPAS2, Serogroup W, Day 0: >=1:4 | 6.8 | 10.8
  PPAS2, Serogroup W, Day 0: >=1:128: number analyzed (Participants) | 148 | 130
  PPAS2, Serogroup W, Day 0: >=1:128 | 0.7 | 0
  PPAS2, Serogroup W, Day 30: >=1:4: number analyzed (Participants) | 171 | 159
  PPAS2, Serogroup W, Day 30: >=1:4 | 100 | 96.9
  PPAS2, Serogroup W, Day 30: >=1:128: number analyzed (Participants) | 171 | 159
  PPAS2, Serogroup W, Day 30: >=1:128 | 90.6 | 56.0
  PPAS3, Serogroup A: >=1:4: number analyzed (Participants) | 103 | 91
  PPAS3, Serogroup A: >=1:4 | 87.4 | 85.7
  PPAS3, Serogroup A: >=1:128: number analyzed (Participants) | 103 | 91
  PPAS3, Serogroup A: >=1:128 | 18.4 | 12.1
  PPAS3, Serogroup C: >=1:4: number analyzed (Participants) | 104 | 94
  PPAS3, Serogroup C: >=1:4 | 99.0 | 77.7
  PPAS3, Serogroup C: >=1:128: number analyzed (Participants) | 104 | 94
  PPAS3, Serogroup C: >=1:128 | 69.2 | 6.4
  PPAS3, Serogroup Y: >=1:4: number analyzed (Participants) | 106 | 93
  PPAS3, Serogroup Y: >=1:4 | 98.1 | 69.9
  PPAS3, Serogroup Y: >=1:128: number analyzed (Participants) | 106 | 93
  PPAS3, Serogroup Y: >=1:128 | 27.4 | 1.1
  PPAS3, Serogroup W: >=1:4: number analyzed (Participants) | 106 | 93
  PPAS3, Serogroup W: >=1:4 | 98.1 | 61.3
  PPAS3, Serogroup W: >=1:128: number analyzed (Participants) | 106 | 93
  PPAS3, Serogroup W: >=1:128 | 33.0 | 3.2

6. Secondary Outcome: Infants Groups 1 and 2: Percentage of Participants With hSBA Antibody Titer >= 4-Fold Rise From Pre-Vaccination to Post-Vaccination
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. Participants with hSBA titers >= 4-fold increase from baseline (pre-vaccination) were analyzed.
Time Frame: PPAS1: At 30 days post first dose (6 to 7 MoA); and PPAS2: At 30 days post second dose (12 to 13 MoA) of MenACYW conjugate vaccine or MENVEO
Population: PPAS1 was a subset of FAS1. FAS1 included all randomized participants who received at least 1 dose of study vaccine in infancy (<12 MOA) and had a valid post vaccination serology result in infancy. PPAS2 was a subset of FAS2. FAS2 included all randomized participants who received at least 1 dose of study vaccine in second year of life (>=12 MOA) and had a valid post vaccination serology result in second year of life. Only participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infants: Group 1 | Infants: Group 2
Number analyzed (Participants) | 143 | 128
percentage of participants
  PPAS1: Serogroup A: number analyzed (Participants) | 108 | 111
  PPAS1: Serogroup A | 30.6 [22.1 to 40.2] | 15.3 [9.2 to 23.4]
  PPAS1: Serogroup C: number analyzed (Participants) | 104 | 107
  PPAS1: Serogroup C | 92.3 [85.4 to 96.6] | 81.3 [72.6 to 88.2]
  PPAS1: Serogroup Y: number analyzed (Participants) | 102 | 106
  PPAS1: Serogroup Y | 30.4 [21.7 to 40.3] | 7.5 [3.3 to 14.3]
  PPAS1: Serogroup W: number analyzed (Participants) | 108 | 112
  PPAS1: Serogroup W | 18.5 [11.7 to 27.1] | 8.0 [3.7 to 14.7]
  PPAS2: Serogroup A: number analyzed (Participants) | 141 | 123
  PPAS2: Serogroup A | 89.4 [83.1 to 93.9] | 82.9 [75.1 to 89.1]
  PPAS2: Serogroup C: number analyzed (Participants) | 134 | 126
  PPAS2: Serogroup C | 99.3 [95.9 to 100] | 97.6 [93.2 to 99.5]
  PPAS2: Serogroup Y: number analyzed (Participants) | 140 | 128
  PPAS2: Serogroup Y | 98.6 [94.9 to 99.8] | 97.7 [93.3 to 99.5]
  PPAS2: Serogroup W: number analyzed (Participants) | 143 | 127
  PPAS2: Serogroup W | 99.3 [96.2 to 100] | 92.9 [87.0 to 96.7]

7. Secondary Outcome: Infants Groups 1 and 2: Percentage of Participants With Vaccine Seroresponse Measured by hSBA at 30 Days Post First Dose of MenACYW Conjugate Vaccine or MENVEO
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. Participants with hSBA vaccine seroresponse which was defined as >= 4-fold increase from baseline (pre-vaccination) were analyzed.
Time Frame: At 30 days post first dose (6 to 7 MoA) of MenACYW conjugate vaccine or MENVEO
Population: The PPAS1 was a subset of the FAS1. The FAS1 included all randomized participants who received at least 1 dose of the study vaccine in infancy (< 12 MOA) and had a valid post vaccination serology result in infancy. Only participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infants: Group 1 | Infants: Group 2
Number analyzed (Participants) | 108 | 112
percentage of participants
  Serogroup A: number analyzed (Participants) | 108 | 111
  Serogroup A | 30.6 [22.1 to 40.2] | 15.3 [9.2 to 23.4]
  Serogroup C: number analyzed (Participants) | 104 | 107
  Serogroup C | 92.3 [85.4 to 96.6] | 81.3 [72.6 to 88.2]
  Serogroup Y: number analyzed (Participants) | 102 | 106
  Serogroup Y | 30.4 [21.7 to 40.3] | 7.5 [3.3 to 14.3]
  Serogroup W | 18.5 [11.7 to 27.1] | 8.0 [3.7 to 14.7]

8. Secondary Outcome: Toddlers Groups 3 and 4: Percentage of Participants With hSBA Antibody Titer >= 1:4 and >= 1:8
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. Participants with hSBA titers >= 1:4 and >= 1:8 were analyzed.
Time Frame: Baseline (Day 0) and 30 days post second dose (20 to 23 MoA) of MenACYW conjugate vaccine or Menactra
Population: The PPAS2 was a subset of the FAS2. The FAS2 included all randomized participants who received at least 1 dose of the study vaccine in the second year of life (>= 12 MOA) and had a valid post vaccination serology result in the second year of life. Only participants with data collected for each specific serogroup at specific timepoint are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Toddlers: Group 3 | Toddlers: Group 4
Number analyzed (Participants) | 61 | 65
percentage of participants
  Serogroup A, Day 0: >=1:4: number analyzed (Participants) | 59 | 59
  Serogroup A, Day 0: >=1:4 | 54.2 [40.8 to 67.3] | 33.9 [22.1 to 47.4]
  Serogroup A, Day 0: >=1:8: number analyzed (Participants) | 59 | 59
  Serogroup A, Day 0: >=1:8 | 28.8 [17.8 to 42.1] | 18.6 [9.7 to 30.9]
  Serogroup A, Day 30: >=1:4: number analyzed (Participants) | 61 | 64
  Serogroup A, Day 30: >=1:4 | 93.4 [84.1 to 98.2] | 76.6 [64.3 to 86.2]
  Serogroup A, Day 30: >=1:8: number analyzed (Participants) | 61 | 64
  Serogroup A, Day 30: >=1:8 | 88.5 [77.8 to 95.3] | 62.5 [49.5 to 74.3]
  Serogroup C, Day 0: >=1:4: number analyzed (Participants) | 59 | 59
  Serogroup C, Day 0: >=1:4 | 3.4 [0.4 to 11.7] | 10.2 [3.8 to 20.8]
  Serogroup C, Day 0: >=1:8: number analyzed (Participants) | 59 | 59
  Serogroup C, Day 0: >=1:8 | 1.7 [0 to 9.1] | 5.1 [1.1 to 14.1]
  Serogroup C, Day 30: >=1:4 | 100 [94.1 to 100] | 98.5 [91.7 to 100]
  Serogroup C, Day 30: >=1:8 | 100 [94.1 to 100] | 98.5 [91.7 to 100]
  Serogroup Y, Day 0: >=1:4: number analyzed (Participants) | 59 | 59
  Serogroup Y, Day 0: >=1:4 | 11.9 [4.9 to 22.9] | 10.2 [3.8 to 20.8]
  Serogroup Y, Day 0: >=1:8: number analyzed (Participants) | 59 | 59
  Serogroup Y, Day 0: >=1:8 | 8.5 [2.8 to 18.7] | 8.5 [2.8 to 18.7]
  Serogroup Y, Day 30: >=1:4 | 100 [94.1 to 100] | 93.8 [85.0 to 98.3]
  Serogroup Y, Day 30: >=1:8 | 100 [94.1 to 100] | 92.3 [83.0 to 97.5]
  Serogroup W, Day 0: >=1:4: number analyzed (Participants) | 59 | 59
  Serogroup W, Day 0: >=1:4 | 1.7 [0 to 9.1] | 3.4 [0.4 to 11.7]
  Serogroup W, Day 0: >=1:8: number analyzed (Participants) | 59 | 59
  Serogroup W, Day 0: >=1:8 | 0 [0 to 6.1] | 1.7 [0 to 9.1]
  Serogroup W, Day 30: >=1:4 | 100 [94.1 to 100] | 86.2 [75.3 to 93.5]
  Serogroup W, Day 30: >=1:8 | 100 [94.1 to 100] | 84.6 [73.5 to 92.4]

9. Secondary Outcome: Toddlers Groups 3 and 4: Geometric Mean Titers Against Meningococcal Serogroups A, C, W, and Y
Description: as for outcome 4
Time Frame: Baseline (Day 0) and 30 days post second dose (20 to 23 MoA) of MenACYW conjugate vaccine or Menactra
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Toddlers: Group 3 | Toddlers: Group 4
Number analyzed (Participants) | 61 | 65
titer
  Serogroup A: Day 0: number analyzed (Participants) | 59 | 59
  Serogroup A: Day 0 | 4.29 [3.36 to 5.49] | 3.43 [2.61 to 4.51]
  Serogroup A: Day 30: number analyzed (Participants) | 61 | 64
  Serogroup A: Day 30 | 45.0 [29.8 to 68.0] | 13.2 [8.72 to 19.9]
  Serogroup C: Day 0: number analyzed (Participants) | 59 | 59
  Serogroup C: Day 0 | 2.10 [1.95 to 2.26] | 2.41 [2.01 to 2.90]
  Serogroup C: Day 30 | 1727 [1300 to 2294] | 59.4 [44.3 to 79.6]
  Serogroup Y: Day 0: number analyzed (Participants) | 59 | 59
  Serogroup Y: Day 0 | 2.44 [2.07 to 2.88] | 2.44 [2.05 to 2.91]
  Serogroup Y: Day 30 | 284 [218 to 369] | 45.5 [32.9 to 62.8]
  Serogroup W: Day 0: number analyzed (Participants) | 59 | 59
  Serogroup W: Day 0 | 2.02 [1.98 to 2.07] | 2.12 [1.93 to 2.34]
  Serogroup W: Day 30 | 202 [152 to 267] | 25.0 [17.6 to 35.7]

10. Secondary Outcome: Toddlers Groups 3 and 4: Percentage of Participants With hSBA Antibody Titer >= 1:4 to >= 1:128
Description: as for outcome 5
Time Frame: Baseline (Day 0) and at 30 days post second dose (20 to 23 MoA) of MenACYW conjugate vaccine or Menactra
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Toddlers: Group 3 | Toddlers: Group 4
Number analyzed (Participants) | 61 | 65
percentage of participants
  Serogroup A, Day 0: >=1:4: number analyzed (Participants) | 59 | 59
  Serogroup A, Day 0: >=1:4 | 54.2 | 33.9
  Serogroup A, Day 0: >=1:128: number analyzed (Participants) | 59 | 59
  Serogroup A, Day 0: >=1:128 | 0 | 3.4
  Serogroup A, Day 30: >=1:4: number analyzed (Participants) | 61 | 64
  Serogroup A, Day 30: >=1:4 | 93.4 | 76.6
  Serogroup A, Day 30: >=1:128: number analyzed (Participants) | 61 | 64
  Serogroup A, Day 30: >=1:128 | 32.8 | 14.1
  Serogroup C, Day 0: >=1:4: number analyzed (Participants) | 59 | 59
  Serogroup C, Day 0: >=1:4 | 3.4 | 10.2
  Serogroup C, Day 0: >=1:128: number analyzed (Participants) | 59 | 59
  Serogroup C, Day 0: >=1:128 | 0 | 1.7
  Serogroup C, Day 30: >=1:4 | 100 | 98.5
  Serogroup C, Day 30: >=1:128 | 100 | 32.3
  Serogroup Y, Day 0: >=1:4: number analyzed (Participants) | 59 | 59
  Serogroup Y, Day 0: >=1:4 | 11.9 | 10.2
  Serogroup Y, Day 0: >=1:128: number analyzed (Participants) | 59 | 59
  Serogroup Y, Day 0: >=1:128 | 0 | 0
  Serogroup Y, Day 30: >=1:4 | 100 | 93.8
  Serogroup Y, Day 30: >=1:128 | 85.2 | 24.6
  Serogroup W, Day 0: >=1:4: number analyzed (Participants) | 59 | 59
  Serogroup W, Day 0: >=1:4 | 1.7 | 3.4
  Serogroup W, Day 0: >=1:128: number analyzed (Participants) | 59 | 59
  Serogroup W, Day 0: >=1:128 | 0 | 0
  Serogroup W, Day 30: >=1:4 | 100 | 86.2
  Serogroup W, Day 30: >=1:128 | 78.7 | 13.8

11. Secondary Outcome: Toddlers Groups 3 and 4: Percentage of Participants With hSBA Antibody Titer >= 4-Fold Rise From Pre-Vaccination to Post-Vaccination
Description: as for outcome 6
Time Frame: At 30 days post second dose (20 to 23 MoA) of MenACYW conjugate vaccine or Menactra
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Toddlers: Group 3 | Toddlers: Group 4
Number analyzed (Participants) | 59 | 59
percentage of participants
  Serogroup A: number analyzed (Participants) | 59 | 58
  Serogroup A | 72.9 [59.7 to 83.6] | 46.6 [33.3 to 60.1]
  Serogroup C | 100 [93.9 to 100] | 93.2 [83.5 to 98.1]
  Serogroup Y | 100 [93.9 to 100] | 88.1 [77.1 to 95.1]
  Serogroup W | 100 [93.9 to 100] | 76.3 [63.4 to 86.4]

12. Secondary Outcome: Toddlers Groups 3 and 4: Percentage of Participants With Vaccine Seroresponse Measured by hSBA at 30 Days Post Second Dose of MenACYW Conjugate Vaccine or Menactra
Description: as for outcome 7
Time Frame: At 30 days post second dose (20 to 23 MoA) of MenACYW conjugate vaccine or Menactra
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Toddlers: Group 3 | Toddlers: Group 4
Number analyzed (Participants) | 59 | 59
percentage of participants
  Serogroup A: number analyzed (Participants) | 59 | 58
  Serogroup A | 72.9 [59.7 to 83.6] | 46.6 [33.3 to 60.1]
  Serogroup C | 100 [93.9 to 100] | 93.2 [83.5 to 98.1]
  Serogroup Y | 100 [93.9 to 100] | 88.1 [77.1 to 95.1]
  Serogroup W | 100 [93.9 to 100] | 76.3 [63.4 to 86.4]

ADVERSE EVENTS:
Time Frame: From the first study vaccine administration (Day 0) up to 6 months after the last vaccination; mean study subject duration was 337 days for groups 1 and 2, and 283 days for groups 3 and 4
Description: Analysis was performed on the overall safety analysis set for any dose.
Arm/Group | Infants: Group 1 | Infants: Group 2 | Toddlers: Group 3 | Toddlers: Group 4
All-Cause Mortality (participants affected / at risk) | 0/370 | 0/361 | 0/96 | 0/103
Serious Adverse Events (participants affected / at risk) | 6/370 | 12/361 | 1/96 | 4/103
Other Adverse Events (participants affected / at risk) | 288/370 | 257/361 | 68/96 | 74/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants: Group 1 (N=370) | Infants: Group 2 (N=361) | Toddlers: Group 3 (N=96) | Toddlers: Group 4 (N=103)
Accidental Exposure To Product (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burns First Degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Croup Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Escherichia Coli (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Parainfluenzae Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal Scalded Skin Syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants: Group 1 (N=370) | Infants: Group 2 (N=361) | Toddlers: Group 3 (N=96) | Toddlers: Group 4 (N=103)
Somnolence (Nervous system disorders) | 160 (208) | 157 (218) | 28 (41) | 30 (36)
Teething (Gastrointestinal disorders) | 29 (44) | 25 (42) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 44 (50) | 39 (41) | 8 (9) | 10 (10)
Decreased Appetite (Metabolism and nutrition disorders) | 83 (104) | 83 (102) | 28 (36) | 34 (47)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 20 (22) | 11 (16) | 1 (1) | 0 (0)
Otitis Media (Infections and infestations) | 15 (17) | 14 (17) | 5 (5) | 5 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 41 (45) | 40 (44) | 3 (4) | 4 (4)
Crying (General disorders) | 160 (200) | 138 (179) | 35 (45) | 34 (45)
Injection Site Bruising (General disorders) | 19 (35) | 13 (17) | 3 (3) | 3 (4)
Injection Site Erythema (General disorders) | 151 (479) | 138 (460) | 29 (41) | 26 (37)
Injection Site Pain (General disorders) | 202 (782) | 180 (691) | 43 (65) | 41 (60)
Injection Site Swelling (General disorders) | 125 (361) | 105 (331) | 23 (34) | 14 (19)
Pyrexia (General disorders) | 68 (83) | 71 (81) | 18 (28) | 20 (23)
Irritability (Psychiatric disorders) | 202 (289) | 186 (264) | 44 (65) | 52 (74)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 6 (8) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03691610/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT03691610/SAP_001.pdf